CLINICAL TRIAL: NCT05806190
Title: Frequency of Nocturnal Hypoglycaemia in Adults With Insulin-treated Diabetes and Adrenal Failure Using Prednisolone or Hydrocortisone: a Pilot Study
Brief Title: Hypoglycaemia (Low Blood Sugar) in Adults With Diabetes and Adrenal Failure
Acronym: HYPO-DIAD
Status: Completed | Type: Observational
Sponsor: Imperial College Healthcare NHS Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 22SM8022
Record Dates: First submitted 2023-03-28; First posted 2023-04-10 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Diabetes Mellitus, Type 1; Adrenal Insufficiency; Diabetes Mellitus Type 2 - Insulin-Treated
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Adrenal Insufficiency | interventions — Continuous Glucose Monitoring

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (2):
- Study group: Participants who live with insulin- treated diabetes and adrenal insufficiency.
  Interventions: Device: Continuous Glucose Monitoring
- Control group: Participants who live with adrenal insufficiency and NOT with insulin-treated diabetes.
  Interventions: Device: Continuous Glucose Monitoring

INTERVENTIONS:
Device: Continuous Glucose Monitoring — Continuous Glucose Monitoring using a Dexcom G6 Continuous Glucose Monitoring Device

SUMMARY:
The purpose of this study is to measure how often low blood sugars occur in people who live with both adrenal insufficiency (AI) and diabetes and need to take insulin. People who live with AI need to take steroid replacement tablets every day, for life. Two of the most common types of steroid replacement tablets are called prednisolone and hydrocortisone.

Low blood sugar (hypoglycemia) is a very common side effect of taking insulin and can often be unpleasant, frightening and dangerous. People who have adrenal failure are also at risk of hypoglycaemia, although this is rare. It is not known whether taking steroids affects how often hypoglycaemia happens.

The study has three aims:

1. To measure how often low blood sugars occur at night in people who live with with both adrenal insufficiency (AI) and insulin-treated diabetes
2. To compare how often low blood sugars occur in people taking prednisolone for their AI versus those taking hydrocortisone.
3. To compare the patterns throughout the day for low blood sugars in those taking prednisolone versus those taking hydrocortisone.

The study will compare this information with results in people who have AI without diabetes.

Participants will be given continuous glucose monitoring systems (Dexcom G6 devices) which are small wearable devices that measure glucose levels throughout the day and night. They will be asked to wear a device for 30 days. Participants will not be asked to make any changes to their usual medications or their diet.

DETAILED DESCRIPTION:
PURPOSE OF THE STUDY

The purpose of this study is to measure how often hypoglycaemia occurs in people who take steroid tablets for adrenal insufficiency and insulin for diabetes compared to individuals with adrenal insufficiency on steroid tablets without diabetes. To do this, participants will be given a continuous glucose monitoring (CGM) system, which is an effective and accurate way of measuring blood sugars throughout the day and night. This study will assess how often hypoglycaemia occurs, especially at night, and whether the type of steroid tablet people take affects how often hypoglycaemia happens.

STUDY AIMS

1. To measure how often low blood sugars occur at night in people with both AI and insulin-treated diabetes using CGM, and in people without diabetes who are matched in age, sex and steroid replacement (hydrocortisone or prednisolone).
2. To compare the frequency of low blood sugars in people taking prednisolone for their AI versus those taking hydrocortisone.
3. To compare the patterns throughout the day for low blood sugars in those taking prednisolone versus those taking hydrocortisone.

STUDY DESIGN

This study will observe 16 adults with both insulin-treated diabetes and adrenal insufficiency and 16 adults without diabetes who are matched for age, sex and steroid replacement. The investigators will aim to recruit 32 participants in total. Participants will spend 30 days in the study.

RECRUITMENT Recruitment will be undertaken in endocrinology and diabetes clinics at Imperial College Healthcare NHS Trust. Participant information sheets will be given to potential participants and following any questions, informed consent will be taken.

Participants will be given as much time as they require (at least 24 hours) to decide whether or not to take part - this can vary on a per participant basis.

ELIGIBILITY:
Inclusion Criteria:

for test group:

* Confirmed diagnoses of adrenal insufficiency and insulin-treated diabetes for more than one year.
* Adults aged above 18 years

for matched control group:

* Diabetes mellitus excluded on baseline blood review
* Adults aged above 18 years

Exclusion Criteria:

* Measured eGFR ≤ 30
* Acute illness
* Abnormal thyroid function
* Admission to hospital
* Pregnant or planning pregnancy
* Breastfeeding
* Enrolled in other clinical trials, except at the discretion of the chief investigator
* Have active malignancy or under investigation for malignancy
* Severe visual impairment
* Reduced manual dexterity
* Unable to participate due to other factors, as assessed by the Chief Investigators

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults living with insulin-treated diabetes and adrenal insufficiency.
Sampling Method: Non-Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2023-04-17 (Actual); Primary Completion 2023-08-31 (Actual); Study Completion 2023-09-15 (Actual)

PRIMARY OUTCOMES:
Time spent in hypoglycaemia | 30 days
  Percentage time spent in hypoglycaemia (glucose levels < 3.0mmol/L, 55mg/dL). Glucose levels will be measured by a continuous glucose monitoring device (CGM).

SECONDARY OUTCOMES:
Time spent in hypoglycaemia (glucose levels < 3.9mmol/L, 70mg/dL) | 30 days
  Percentage time spent in hypoglycaemia (glucose levels < 3.9mmol/L, 70mg/dL)
Time spent in target glucose levels | 30 days
  Percentage time spent in target (glucose levels 3.9-10mmol/L, 70-180mg/dL)
Time spent in hyperglycaemia | 30 days
  Percentage time spent in hyperglycaemia (glucose levels >10mmol/L, 180mg/dL)
Hypoglycaemic excursions | 30 days
  Number of hyperglycaemic excursions. This will comprise the number of times glucose sugar levels are recorded as below 3.9mmol/L, 70mg/dL
Gold questionnaire score | Baseline
  The Gold questionnaire asks individuals to report their experience in detecting hypoglycemic events with scores ranging from minimum score of 1 (always aware) to a maximum score of 7 (never aware). The minimum score refers to the individual never being aware of hypoglycaemia, and an increasing score refers to greater awareness of hypoglycaemia.
Hypoglycaemia Fear Survey-II (HFS-II) score | Baseline
  This 33-item questionnaire assesses fear of hypoglycaemia. The minimum score is 0 and the maximum score is 132. A higher score indicated greater fear of hypoglycaemia.
Hospital Anxiety and Depression (HADS) Score | Baseline
  A questionnaire assessing levels of anxiety and depression. The questionnaire consists of 14 questions: 7 questions assess for anxiety and 7 questions assess for depression. Each question can score between 0 and 3. Two scores are calculated separately for anxiety and depression. The minimum score is 0 and maximum score is 21 for both anxiety and depression. A greater score denotes greater severity of anxiety or depression.

CONTACTS AND LOCATIONS:
Locations (1):
- Charing Cross Hospital, Imperial College Healthcare NHS Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bensing S, Brandt L, Tabaroj F, Sjoberg O, Nilsson B, Ekbom A, Blomqvist P, Kampe O. Increased death risk and altered cancer incidence pattern in patients with isolated or combined autoimmune primary adrenocortical insufficiency. Clin Endocrinol (Oxf). 2008 Nov;69(5):697-704. doi: 10.1111/j.1365-2265.2008.03340.x. Epub 2008 Aug 22. PMID 18727712
- [Background] Bergthorsdottir R, Leonsson-Zachrisson M, Oden A, Johannsson G. Premature mortality in patients with Addison's disease: a population-based study. J Clin Endocrinol Metab. 2006 Dec;91(12):4849-53. doi: 10.1210/jc.2006-0076. Epub 2006 Sep 12. PMID 16968806
- [Background] Chantzichristos D, Persson A, Eliasson B, Miftaraj M, Franzen S, Bergthorsdottir R, Gudbjornsdottir S, Svensson AM, Johannsson G. Mortality in patients with diabetes mellitus and Addison's disease: a nationwide, matched, observational cohort study. Eur J Endocrinol. 2017 Jan;176(1):31-39. doi: 10.1530/EJE-16-0657. PMID 27928991
- [Background] Julious SA. Sample size of 12 per group rule of thumb for a pilot study. Pharmaceutical Statistics. 2005;4(4):287-291. doi:https://doi.org/10.1002/pst.185
- [Background] Lu CL, Shen HN, Hu SC, Wang JD, Li CY. A Population-Based Study of All-Cause Mortality and Cardiovascular Disease in Association With Prior History of Hypoglycemia Among Patients With Type 1 Diabetes. Diabetes Care. 2016 Sep;39(9):1571-8. doi: 10.2337/dc15-2418. Epub 2016 Jul 6. PMID 27385329
- [Background] Ngaosuwan K, Johnston DG, Godsland IF, Cox J, Majeed A, Quint JK, Oliver N, Robinson S. Cardiovascular Disease in Patients With Primary and Secondary Adrenal Insufficiency and the Role of Comorbidities. J Clin Endocrinol Metab. 2021 Apr 23;106(5):1284-1293. doi: 10.1210/clinem/dgab063. PMID 33585930
- [Background] Ngaosuwan K, Johnston DG, Godsland IF, Cox J, Majeed A, Quint JK, Oliver N, Robinson S. Increased Mortality Risk in Patients With Primary and Secondary Adrenal Insufficiency. J Clin Endocrinol Metab. 2021 Jun 16;106(7):e2759-e2768. doi: 10.1210/clinem/dgab096. PMID 33596308
- [Background] Ngaosuwan K, Johnston DG, Godsland IF, Cox J, Majeed A, Quint JK, Oliver N, Robinson S. Mortality Risk in Patients With Adrenal Insufficiency Using Prednisolone or Hydrocortisone: A Retrospective Cohort Study. J Clin Endocrinol Metab. 2021 Jul 13;106(8):2242-2251. doi: 10.1210/clinem/dgab347. PMID 33993277
- [Background] Rao Kondapally Seshasai S, Kaptoge S, Thompson A, Di Angelantonio E, Gao P, Sarwar N, Whincup PH, Mukamal KJ, Gillum RF, Holme I, Njolstad I, Fletcher A, Nilsson P, Lewington S, Collins R, Gudnason V, Thompson SG, Sattar N, Selvin E, Hu FB, Danesh J; Emerging Risk Factors Collaboration. Diabetes mellitus, fasting glucose, and risk of cause-specific death. N Engl J Med. 2011 Mar 3;364(9):829-841. doi: 10.1056/NEJMoa1008862. PMID 21366474
- [Background] Emerging Risk Factors Collaboration; Sarwar N, Gao P, Seshasai SR, Gobin R, Kaptoge S, Di Angelantonio E, Ingelsson E, Lawlor DA, Selvin E, Stampfer M, Stehouwer CD, Lewington S, Pennells L, Thompson A, Sattar N, White IR, Ray KK, Danesh J. Diabetes mellitus, fasting blood glucose concentration, and risk of vascular disease: a collaborative meta-analysis of 102 prospective studies. Lancet. 2010 Jun 26;375(9733):2215-22. doi: 10.1016/S0140-6736(10)60484-9. PMID 20609967

DOCUMENTS (2):
  • Study Protocol (2023-03-09): https://cdn.clinicaltrials.gov/large-docs/90/NCT05806190/Prot_000.pdf
  • Informed Consent Form (2023-03-08): https://cdn.clinicaltrials.gov/large-docs/90/NCT05806190/ICF_001.pdf